CLINICAL TRIAL: NCT00322660
Title: Can the Risk of RD and Hypoglycemia in Children Born at Elective CS be Reduced by Injection of Adrenaline
Brief Title: Adrenaline Injections to Children Born at Elective CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2005091
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Respiratory Distress; Hypoglycemia
MeSH Terms: conditions — Dyspnea; Hypoglycemia | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Adrenaline

SUMMARY:
Children born after elective C-section have a greater risk of respiratory problems and hypoglycemia - most likely due to a lower concentration of stress hormones compared to children born vaginally. Hypothesis: can we eliminate or reduce the risk of respiratory distress and hypoglycaemia by administrating adrenaline to the newborn.

ELIGIBILITY:
Inclusion Criteria:

* All children born at elective section with gestational age more than 37 + 0

Exclusion Criteria:

* Children in whom a serious malformation was found during pregnancy assuming this malformation will lead to very early death or respiratory problems.
* Serious malformations (ex.anencephalia) will be excluded at birth
* Other malformations will be estimated by investigator whether it will lead to exclusion.

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2006-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
respiratory distress
hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Lene A Olsen, M.D., Principal Investigator — Hvidovre University Hospital, Copenhagen, Kettegaards allé 30, 2650 Hvidovre, DK; Pernille Pedersen, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Copenhagen, Hvidovre
  - Hvidovre Hospital, Kettegård Alle 31, Hvidovre

REFERENCES:
- [Background] Irestedt L, Lagercrantz H, Belfrage P. Causes and consequences of maternal and fetal sympathoadrenal activation during parturition. Acta Obstet Gynecol Scand Suppl. 1984;118:111-5. doi: 10.3109/00016348409157136. PMID 6587720
- [Derived] Pedersen P, Avlund OL, Pedersen BL, Pryds O. Intramuscular adrenaline does not reduce the incidence of respiratory distress and hypoglycaemia in neonates delivered by elective caesarean section at term. Arch Dis Child Fetal Neonatal Ed. 2009 May;94(3):F164-7. doi: 10.1136/adc.2008.138487. Epub 2008 Sep 11. PMID 18786961